CLINICAL TRIAL: NCT00099125
Title: A Phase II Study Of Radiation Therapy Plus Low Dose Temozolomide Followed By Temozolomide Plus Irinotecan For Glioblastoma Multiforme
Brief Title: Radiation Therapy, Temozolomide, and Irinotecan in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0420; CDR0000389229
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult gliosarcoma; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Irinotecan; Temozolomide; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RT with chemotherapy + post-radiation chemotherapy (Experimental): Radiation therapy (RT) with concurrent chemotherapy + post-radiation chemotherapy
  Interventions: Drug: irinotecan hydrochloride; Drug: temozolomide; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: temozolomide
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy, such as temozolomide and irinotecan, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well radiation therapy, temozolomide, and irinotecan work in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall survival of patients with newly diagnosed supratentorial glioblastoma multiforme treated with radiotherapy and temozolomide followed by temozolomide and irinotecan with historical controls from the RTOG database.
* Determine the short- and long-term toxicity of this regimen in these patients.
* Determine progression-free survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Chemoradiotherapy: Patients undergo radiotherapy once daily, 5 days a week, for 6 weeks. Concurrently with radiotherapy, patients receive oral temozolomide once daily, 7 days a week, for 6 weeks.
* Post-radiotherapy chemotherapy: Beginning 4-6 weeks after the completion of chemoradiotherapy, patients receive irinotecan IV on days 1 and 15 and oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 157 patients will be accrued for this study within 11 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed supratentorial glioblastoma multiforme by surgical biopsy or excision

  * No gliomas graded less than glioblastoma multiforme
  * No recurrent malignant gliomas
* No tumor foci below the tentorium or beyond the cranial vault
* Study therapy must begin ≤ 5 weeks after surgery

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* At least 8 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL*
* Hematocrit ≥ 30%* NOTE: *Transfusion allowed

Hepatic

* Bilirubin ≤ 0.5 mg/dL
* ALT or AST ≤ 2 times upper limit of normal

Renal

* Creatinine ≤ 1.5 mg/dL
* BUN ≤ 25 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception during and for 2 months after study participation
* No AIDS
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix or bladder
* No other major medical illness or psychiatric impairment that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent sargramostim (GM-CSF)

Chemotherapy

* No other concurrent chemotherapy

Endocrine therapy

* Concurrent steroid therapy allowed provided patient is on a stable or decreasing dose for at least 2 weeks before study entry

Radiotherapy

* No prior radiotherapy to the head or neck resulting in overlap of radiotherapy fields

  * Prior radiotherapy for stage T1 glottic cancer allowed

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Other

* No enzyme-inducing antiepileptic drugs within 14 days before the initiation of irinotecan

  * Concurrent non-enzyme-inducing antiepileptic drugs allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2004-11; Primary Completion 2006-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | From registration to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 18 months.

SECONDARY OUTCOMES:
Progression-free survival | From randomization to date of progression, death, or last follow-up. Analysis occurs at the same time as the primary outcome analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Frank S. Lieberman, MD, Study Chair — University of Pittsburgh; Christina I. Tsien, MD, Study Chair — University of Michigan Rogel Cancer Center
Locations (118):
- United States (118):
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Saint Agnes Medical Center, Fresno, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Providence Holy Cross Cancer Center, Mission Hills, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Radiological Associates of Sacramento Medical Group, Inc., Sacramento, California
  - Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Tulane Cancer Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Cancer Institute of Cape Girardeau, Cape Girardeau, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Dartmouth - Hitchcock Concord, Concord, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - Cooper Cancer Institute, Camden, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - John Smith, Jr./Dalton McMichael Cancer Center at Morehead Memorial Hospital, Eden, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Akron City Hospital, Akron, Ohio
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Radiation Oncology Center, Alliance, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Glesham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Comprehensive Cancer Center at Legacy Good Samaritan Hospital & Medical Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Cancer Center - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UPMC McKeesport, McKeesport, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC - Shadyside, Pittsburgh, Pennsylvania
  - UPMC - Passavant Hospital, Pittsburgh, Pennsylvania
  - Cancer Center at St. Clair Memorial Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Wellspan Health, York, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Community Cancer Center at Rutland Regional Medical Center, Rutland, Vermont
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - North Star Lodge Cancer Center, Yakima, Washington
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Lieberman FS, Tsien C, Berkey B, et al.: Phase II trial of concomitant low dose temozolomide with external beam radiation (EBRT) followed by 12 months of temozolomide and irinotecan for newly diagnosed glioblastoma (GBM): preliminary results of RTOG 04-20. [Abstract] J Clin Oncol 24 (Suppl 18): A-1510, 2006.